CLINICAL TRIAL: NCT01848782
Title: Impact of Adding a Limitation Section in Abstract of Systematic Review on Interpretation by Readers: a Randomised Controlled Trial
Brief Title: Impact of Adding a Limitation Section in Abstract of Systematic Review
Acronym: ILMARI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RAV006
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2013-04

CONDITIONS: Systematic Review
Keywords: abstract; meta-analysis; systematic review; interpretation; results; quality; bias; spin; limits; limitation; risk of bias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- abstract with limitation section added (Experimental): we add a limitation section in each selected abstract, the limitation section will focus on the quality of included studies.
  Interventions: Behavioral: interpretation of the abstract of the systematic review
- abstract without limitation section (Active Comparator): We selected 30 abstracts with a conclusion in favour the experimental treatment from a sample of systematic reviews that evaluate the effect of health care intervention.
  Interventions: Behavioral: interpretation of the abstract of the systematic review

INTERVENTIONS:
Behavioral: interpretation of the abstract of the systematic review

SUMMARY:
Objective: The investigators aim to evaluate the impact of a adding a " limitations " section in systematic review's abstract on result's interpretation by readers Design: randomized controlled trial with two parallel arms. Participants will be invited to participate in an online survey.

Participants: Eligible participants are corresponding authors of clinical trials published between 2010 and 2012 and referenced in Medline.

Intervention: The investigators will evaluate the impact of the presence of a " limitations " section in abstract of systematic review with meta- analysis. The investigators selected abstracts of meta-analysis from a sample.

Selected abstract will be standardised and the treatment's name hidden. Two groups of abstract will be presented as follow: 1) abstract without " limitations " section 2) abstract with " limitations " section. The " limitations " section will be written by authors and will briefly describe the risk of bias of included studies.

Selected participant are invited by e-mail to answer the survey. After reading one abstract from his/her group of randomisation they are invited to answer 5 questions about their interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

* corresponding authors of clinical trail indexed in pubmed with email address available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amelie YAVCHITZ, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Yavchitz A, Ravaud P, Hopewell S, Baron G, Boutron I. Impact of adding a limitations section to abstracts of systematic reviews on readers' interpretation: a randomized controlled trial. BMC Med Res Methodol. 2014 Nov 24;14:123. doi: 10.1186/1471-2288-14-123. PMID 25420433

RESULTS

PARTICIPANT FLOW:
Groups:
- Abstract With Limitation Section Added: we add a limitation section in each selected abstract, the limitation section will focus on the quality of included studies.
  interpretation of the abstract of the systematic review
- Abstract Without Limitation Section: We selected 30 abstracts with a conclusion in favour the experimental treatment from a sample of systematic reviews that evaluate the effect of health care intervention.
  interpretation of the abstract of the systematic review
Period: Overall Study
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.3) | 46.7 (10.9) | 46.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 109 | 107 | 216
Education qualification [Count of Participants; unit: Participants]
  MD | 78 | 78 | 156
  PhD | 58 | 64 | 122
  Other | 14 | 8 | 22
Clinical experience [Count of Participants; unit: Participants]
  <5 years | 6 | 8 | 14
  5 to 10 years | 34 | 28 | 62
  >10 years | 110 | 114 | 224
Reading reports of systematic reviews [Count of Participants; unit: Participants]
  Rarely or sometimes | 61 | 62 | 123
  Regularly | 89 | 87 | 176
No. of randomized trials involved in [Count of Participants; unit: Participants]
  0 trial | 16 | 11 | 27
  1-3 trials | 48 | 48 | 96
  4-9 trials | 45 | 54 | 99
  >10 trials | 41 | 37 | 78
Authored at least one systematic review [Count of Participants; unit: Participants] | 77 | 82 | 159
No. of systematic reviews peer-reviewed [Count of Participants; unit: Participants]
  0 review | 75 | 64 | 139
  1-3 reviews | 55 | 69 | 124
  >3 reviews | 20 | 16 | 36
Training in clinical epidemiology [Count of Participants; unit: Participants] | 101 | 76 | 177
Training in methods of randomized trials [Count of Participants; unit: Participants] | 86 | 71 | 157

OUTCOME MEASURES:

1. Primary Outcome: Confidence in the Results of the Systematic Review
Description: we ask participants: "how confident are you in the results of this study?", with the choice of answer based on a 10 points Likert scale (score from 0, not at all confident, to 10, very confident )
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Number analyzed (Participants) | 150 | 150
score on a scale | 4.6 (2.5) | 4.4 (2.3)
Statistical Analysis 1: Comparison: Abstract With Limitation Section Added vs Abstract Without Limitation Section; Test type: Superiority; p = 0.5, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.7]

2. Secondary Outcome: Confidence With the Validity of the Conclusions
Description: We ask participants:
  - "How confident are you in the validity of the conclusions of this study?"
  with the choice of answer based on a 10 points Likert scale from 0, not at all confident, to 10, very confident
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Number analyzed (Participants) | 150 | 150
score on a scale | 4.1 (2.5) | 4.0 (2.3)
Statistical Analysis 1: Comparison: Abstract With Limitation Section Added vs Abstract Without Limitation Section; Test type: Superiority; p = 0.8, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.5 to 0.6]

3. Secondary Outcome: Beneficial Effect of the Experimental Intervention
Description: We ask participants:
  - "How confident are you that the intervention "A" could be of benefit to patients?"
  with the choice of answer based on a 10 points Likert scale from 0, not at all confident, to 10, very confident
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Number analyzed (Participants) | 150 | 150
score on a scale | 4.4 (2.6) | 4.3 (2.3)
Statistical Analysis 1: Comparison: Abstract With Limitation Section Added vs Abstract Without Limitation Section; Test type: Superiority; p = 0.6, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.7]

4. Secondary Outcome: Influence of Results on Clinical Practice
Description: We ask participants:
  "How confident are you that the results of this study could influence your clinical practice?" with the choice of answer based on a 10 points Likert scale from 0, not at all confident, to 10, very confident
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Number analyzed (Participants) | 150 | 150
score on a scale | 3.8 (2.6) | 3.8 (2.3)
Statistical Analysis 1: Comparison: Abstract With Limitation Section Added vs Abstract Without Limitation Section; Test type: Superiority; p = 0.8, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.6 to 0.5]

5. Secondary Outcome: The Rigor of the Systematic Review
Description: We ask participants:
  "Do you think that this systematic review was conducted rigorously?" with the choice of answer based on a 10 points Likert scale from 0, not at all confident, to 10, very confident
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
Number analyzed (Participants) | 150 | 150
score on a scale | 4.1 (2.7) | 4.4 (2.6)
Statistical Analysis 1: Comparison: Abstract With Limitation Section Added vs Abstract Without Limitation Section; Test type: Superiority; p = 0.2, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.0 to 0.2]

ADVERSE EVENTS:
Arm/Group | Abstract With Limitation Section Added | Abstract Without Limitation Section
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No